CLINICAL TRIAL: NCT04978467
Title: Feasibility of Using Maestro Hand Exoskeleton in Post-stroke Hand Rehabilitation to Improve Joint Coordination
Brief Title: SPiRE Maestro Hand Exoskeleton for Rehabilitation Post Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Device implementation delayed
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3869-P
Record Dates: First submitted 2021-07-16; First posted 2021-07-27 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: Soft Robotics; Robotic Exoskeleton; Neurologic Rehabilitation; Physical Medicine and Rehabilitation; Rehabilitation Exercise
MeSH Terms: conditions — Stroke | interventions — Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: All participants will experience all controller conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental): All participants will receive assistance to move finger joints away from the compensatory coordination (compensation avoidance), toward the desired trajectories (task assistance), both, and none in different days.
  Interventions: Device: Exoskeleton

INTERVENTIONS:
Device: Exoskeleton — Participants will receive assistance to move finger joints away from the compensatory coordination (compensation avoidance), toward the desired trajectories (task assistance), both, and none in different days.

SUMMARY:
The research team will develop a novel training tool to improve finger joint coordination, to address the unmet need in the current rehabilitation, thereby enhancing hand function and contributing to improved independence and quality of life for Veterans with stroke.

DETAILED DESCRIPTION:
The research team will determine feasibility of training using CA and TA controllers in subacute stroke. Specifically, we will examine if joint coordination improves over a training session. The investigators will compare the extent of improvement for each controller and impairment severity.

ELIGIBILITY:
Inclusion Criteria:

* Adult Veterans with a stroke 1-6 months ago
* Ability to move fingers (Chedoke-McMaster Hand Section Stage 2-4)

Exclusion Criteria:

* Inability to follow 2-step commands
* Severe muscle tone prohibiting proper placement of the fingers (Modified Ashworth Scale, MAS=5 out of 5)
* Change in spasticity medication or botulinum toxin injection in the upper limb within 3 months prior to or during enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
change in finger joint torque assistance | from the 1st half to the 2nd half of the 1-hour training session
  Change in finger joint torque assistance needed from the 1st half to the 2nd half of the 1-hour training session. Reduction in torque is considered a good outcome. There is no predefined minimum/maximum.

CONTACTS AND LOCATIONS:
Overall Officials: Na Jin Seo, PhD MS BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Due to the small sample size, individual data that are de-identified will be presented in publications.
Time Frame: De-identified individual data that are presented in publications will be available as long as the publications are available.
Access Criteria: Journals' access criteria.